CLINICAL TRIAL: NCT05724173
Title: Single Neuron Population Dynamics in Human Speech Motor Cortex for a Speech Prosthesis
Brief Title: Feasibility of the BrainGate2 Neural Interface System in Persons With Tetraplegia
Acronym: BG-Speech-01
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Leigh R. Hochberg, MD, PhD. (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor-Investigator, Leigh R. Hochberg, MD, PhD., Neurologist, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022p003220 (BG-Speech-01); U01DC019430 (NIH)
Record Dates: First submitted 2023-01-12; First posted 2023-02-13 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Anarthria; Dysarthria; Tetraplegia; Spinal Cord Injuries; Amyotrophic Lateral Sclerosis; Brain Stem Infarctions; Locked in Syndrome; Muscular Dystrophies
MeSH Terms: conditions — Dysarthria; Quadriplegia; Spinal Cord Injuries; Amyotrophic Lateral Sclerosis; Brain Stem Infarctions; Locked-In Syndrome; Muscular Dystrophies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- BrainGate Neural Interface System (Other): Placement of the BrainGate2 sensor(s) into the speech-related cortex
  Interventions: Device: BrainGate Neural Interface System

INTERVENTIONS:
Device: BrainGate Neural Interface System — Placement of the BrainGate2 sensor(s) into the speech-related cortex

SUMMARY:
The purpose of this study is to obtain preliminary device safety information and demonstrate proof of principle (feasibility) of the ability of people with tetraplegia to control a computer cursor and other assistive devices with their thoughts.

DETAILED DESCRIPTION:
The goal of the BrainGate2 research and development project is to identify the core methods and features for a medical device that could allow people with paralysis, including severe speech impairment, to recover a host of abilities that normally rely on the hands or on speech.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 80 years of age.
* Participants must have a diagnosis of amyotrophic lateral sclerosis (ALS) as verified by a clinical expert in neurologic diseases.
* Participants with a diagnosis of ALS with anarthria, or severe dysarthria with decline in the preceding four months.
* Must be within a three-hour drive of the Study site and geographically stable for at least 15 months after enrollment.

Exclusion Criteria:

* Visual impairment such that extended viewing of a computer monitor would be difficult even with ordinary corrective lenses
* Chronic oral or intravenous steroids or immunosuppressive therapy
* Other serious disease or disorder that could seriously affect ability to participate in the study

(There are additional exclusion criteria)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Device Safety | 1 year
  To determine the safety of the Sensor and overall safety of the System. Participants will be considered a success for this safety measure if they are successfully implanted with the Sensor(s) and:
  1. the sensors are not explanted for safety reasons during the one-year post-implant evaluation period.
  2. there are no device-related Serious Adverse Events that result in death or permanently increased disability during the one-year post-implant evaluation period.

SECONDARY OUTCOMES:
Device Feasibility | At participant exit from study, or up to 5 years
  The purpose of this feasibility measure is to define the metrics by which a larger trial of intracortical recording for the restoration of speech-based communication might be planned.
  The secondary endpoints are:
  Number of participants that are able to use the BrainGate system to communicate via speech decoding:
  1. at a rate of at least 5 words per minute and
  2. with less than a median word error rate of 50%.

CONTACTS AND LOCATIONS:
Overall Officials: Jaimie Henderson, MD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Stanford University School of Medicine, Stanford, California
  - Massachusetts General Hospital, Boston, Massachusetts